CLINICAL TRIAL: NCT06687733
Title: A Phase I/II Study for the Safety and Efficacy of Intravenous Infusion With NGGT002 in Adults Patients With Classic Phenylketonuria
Brief Title: Safety and Efficacy Study of NGGT002 in cPKU Adult Subjects
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NGGT (Suzhou) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGGT002-P-2302
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGGT002 (Experimental): Six to eighteen patients will be enrolled into three cohorts at three dose levels.
  Interventions: Genetic: NGGT002

INTERVENTIONS:
Genetic: NGGT002 — adeno-associated viral vector with human phenylalanine hydroxylase gene

SUMMARY:
This is a Phase 1/2, open-label, multiple-center, dose escalation and cohort expansion study to evaluate the safety and efficacy of NGGT002 in adult subjects with classic Phenylketonuria (PKU). NGGT002 is a rAAV8 based vector carrying a functional copy of the human PAH gene.

Participants will receive a single administration of NGGT002 and will be followed for safety and efficacy for 5 years.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of NGGT002 gene therapy with three dose cohorts in adult subjects with a diagnosis of classic PKU, a condition characterized by severe PAH deficiency with no residual enzyme activity. NGGT002 will be administered through intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participating in the study and signing the informed consent form;
2. Gender is not limited; patients must carry biallelic pathogenic or likely pathogenic variants in the PAH gene;
3. Adult patients aged 18 to 55 years;
4. In the past 24 months, at least two blood Phe concentrations have been ≥600 μmol/L (10 mg/dL), with at least one of these measurements taken within 6 months prior to the screening period;
5. Willing and able to manage their diet;
6. According to the investigator's opinion, willing and able to comply with the study procedures and requirements;
7. Women of childbearing potential must have a negative serum HCG test within 7 days before dosing. Participants must agree to use highly effective contraceptive measures for at least one year after receiving NGGT002.

Exclusion Criteria:

1. Presence of anti-AAV8 neutralizing antibodies（≥1:5）
2. Subjects whose disease is well-controlled with existing therapies, such as those currently receiving medications like Sapropterin Dihydrochloride tablets, Pegvaliase-pqpz, etc.;
3. Before dosing, the patient's hematological laboratory tests exceed any of the following limits:

   * Alanine Transaminase (ALT) > 1.5×ULN and/or Aspartate Aminotransferase (AST) > 1.5×ULN
   * Alkaline Phosphatase (ALP) > 1.5×ULN
   * Total Bilirubin (TBil) > 1.5×ULN, Direct Bilirubin > 1.5×ULN
   * International Normalized Ratio (INR) > 1.5
   * Serum Creatinine (Scr) > 1.5×ULN
   * Hematological values outside the normal range (Hemoglobin: <110 g/L for males, <100 g/L for females, White Blood Cells <3.0×10^9/L, Neutrophils <1.5×10^9/L, Platelets <100×10^9/L)
   * Glycated Hemoglobin (HbA1c) > 6% or Fasting Blood Glucose > 6.1 mmol/L
4. At screening, clinically significant abnormal vital signs, physical examination, laboratory test results, or other relevant findings that, in the investigator's opinion, make the subject unsuitable for inclusion;
5. In the investigator's assessment, the subject has contraindications to corticosteroid use or conditions that could lead to a worsening of the condition;
6. Hepatitis A virus infection, active or occult hepatitis B virus infection, active hepatitis C virus infection, positive for Human Immunodeficiency Virus (HIV) antibodies, positive syphilis test, active or latent tuberculosis (TB) infection;
7. A significant history of liver disease, such as steatosis, fibrosis, non-alcoholic steatohepatitis, and cirrhosis, biliary diseases, within 6 months prior to signing the informed consent form, except for Gilbert's syndrome;
8. History of malignant tumors;
9. Imaging (liver ultrasound) evidence of severe liver diseases such as hepatic fibrosis or cirrhosis;
10. In the investigator's assessment, the subject has a history of serious cardiovascular, respiratory, gastrointestinal, endocrine, renal, hematological, neurological, psychiatric, or other systemic diseases before screening;
11. History of allergy to human serum albumin;
12. Subjects with a history of substance abuse (e.g., alcohol, heroin, amphetamines, etc.);
13. Subjects who have received gene therapy at any time in the past.
14. Subjects who have participated in other non-gene therapy drug clinical trials and received the investigational drug within 3 months (or 5 half-lives of the other investigational drug) prior to screening;
15. Subjects with elevated Alpha-fetoprotein (AFP);
16. Other conditions that, in the investigator's opinion, make the subject unsuitable for inclusion, such as severe comorbidities associated with PKU (e.g., renal insufficiency or renal failure, osteoporosis, anemia, gastroesophageal reflux or peptic ulcer, major depressive disorder, epilepsy, etc.);
17. Subjects weighing more than 100 kg;
18. Subjects whose daily diet includes excessive natural protein intake (>2 g/kg/day).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | Baseline to Week 52
  Incidence and severity of AEs, including serious AEs (SAEs) as assessed by CTCAE v5.0 of a single administration of NGGT002.
Change from baseline in average Plasma Phe Concentration | Week 12, Week 28, Week 52
  To evaluate the efficacy in change of average plasma Phe concentration of IV infusion of NGGT002 in adults with classic PKU at Week 12, Week 28, Week 52

SECONDARY OUTCOMES:
Incidence of sustained plasma Phe concentration of ≤360 μmol/L (6 mg/dL) at Week 12, Week 28, Week 52 post dose | Week 12, Week 28, Week 52
  Subjects achieving a sustained plasma Phe concentration ≤360 μmol/L (6 mg/dL) at Week 12, Week 28, Week 52 post dose.
Occurred Day to first reach Phe ≤ 360 μmol/L and the duration（days） of Phe ≤ 360 μmol/L in each dose group following NGGT002 administration | Week 52
  Time（days） to first reach Phe ≤ 360 μmol/L and the duration（days） of Phe ≤ 360 μmol/L in each dose group following NGGT002 administration
Change from baseline in Phe and total protein intake at Week 28, Week 52 post dose | Week 28, Week 52
  Subject achieving a change from baseline in Phe and total protein intake at Week 28, Week 52 post dose.
Score change in Phenylketonuria Quality of Life Questionnaire (PKU-QOL) | Week 28, Week 52
  Score change in PKU-QOL at Week 28, Week 52 post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Weng, PhD, Principal Investigator — First Affiliated Hospital of Bengbu Medical College
Locations (2):
- China (2):
  - First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Xinhua Hospital Affifiated to Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No